CLINICAL TRIAL: NCT00578006
Title: Pilot Study of STAR, an Internet-based System for Cancer Patients to Self-report Toxicity Symptoms, Performance Status, and Quality of Life
Brief Title: Internet-based System for Cancer Patients to Self-report Toxicity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 04-020
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Cervical Cancer; Lung Cancer; Prostate Cancer; Vaginal Cancer; Ovarian Cancer; Breast Cancer; Bladder Cancer
Keywords: toxicity related symptoms; 04-020
MeSH Terms: conditions — Uterine Cervical Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Vaginal Neoplasms; Ovarian Neoplasms; Breast Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): If you are in group A, the investigators will ask you to fill out a brief paper questionnaire periodically to tell us how you are feeling, and how satisfied you are with your care.
  Interventions: Behavioral: Questioners
- B (Experimental): If you are in group B, the investigators will provide you with access to the STAR website using a computer in the waiting area, into which you can report your symptoms every time you come to Sloan-Kettering for an appointment or chemotherapy. The investigators may also provide you with a website address so that you can access STAR from home (or any other location) to report your symptoms at any time.
  Interventions: Behavioral: STAR website

INTERVENTIONS:
Behavioral: Questioners — The investigators will ask you to fill out a brief paper questionnaire periodically to tell us how you are feeling, and how satisfied you are with your care.
  Arms: A
Behavioral: STAR website — You can report your symptoms every time you come to Sloan-Kettering for an appointment or chemotherapy.
  Arms: B

SUMMARY:
Cancer patients may develop side effects during treatment, such as nausea, pain, fatigue, diarrhea, constipation, or shortness of breath. These symptoms may be due to the cancer itself, or due to treatments like chemotherapy drugs or radiation therapy. Doctors and nurses often ask patients about their symptoms, because an important part of cancer treatment is to make patients feel as well as possible. If patients do not feel well, the investigators may need to change the way the investigators are treating you or prescribe therapies that will decrease your symptoms. The best way to find out how you are feeling is to ask you directly.

However, during your time between appointments the investigators may not be able to ask you how you are feeling on a regular basis. In addition, even at an appointment, there may be symptoms that the investigators do not have a chance to discuss.

The investigators are interested in developing new ways to ask patients about how they are feeling, using the Internet. A special new website called STAR ("Symptom Tracking and Reporting for Patients") has been developed to help patients record this information, so that their doctors and nurses can review it during clinic appointments. This study is designed to help us see if STAR is a helpful way for us to keep track of information about patients' symptoms and quality of life.

DETAILED DESCRIPTION:
This pilot study will assess patient use of STAR (Symptom Tracking and Reporting for Patients), an online system designed for cancer patients to self-record toxicity-related symptoms based on NCI Common Terminology Criteria for Adverse Events v3.0, performance status by ECOG criteria, global quality of life by the EuroQOL 5-D assessment tool, emergency room visits, and survival. Secondary outcomes will include patient assessment of the usefulness of STAR, clinician perceptions of the potential value of STAR in routine clinical practice, and an evaluation of whether STAR improves the patient experience of care as assessed by satisfaction measures.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Diagnosis of gynecologic (ovarian; cervical; uterine; primary peritoneal), lung (non-small cell; small cell), gastrointestinal (colorectal, rectal, gastric, esophageal, GI neuroendocrine, small intestine malignancy, pancreatic, hepatocellular), breast, bladder cancer or prostate malignancy
* Receiving primary medical oncology care at MSKCC medical oncology outpatient clinics
* Receiving cytotoxic chemotherapy not on a clinical trial (or a new hormonal therapy in the case of prostate cancer patients only), with treatment expected to continue for at least four weeks from the time of enrollment
* Signed informed consent and Research Authorization

Exclusion Criteria:

* ECOG performance status greater than 2
* Unable to read and comprehend English language text

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1007 (Actual)
Dates: Start 2004-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
To evaluate patient willingness to use STAR (Symptom Tracking and Reporting for Patients), an Internet-based system for cancer patients to self-report common toxicity symptoms, performance status, and quality of life. | conclusion of study
To evaluate the impact of STAR on clinical outcomes | 2 years

SECONDARY OUTCOMES:
To measure patient assessments of the usefulness of STAR, and to measure clinician perceptions of the potential value of STAR in routine outpatient cancer care. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Ethan Basch, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Basch E, Deal AM, Kris MG, Scher HI, Hudis CA, Sabbatini P, Rogak L, Bennett AV, Dueck AC, Atkinson TM, Chou JF, Dulko D, Sit L, Barz A, Novotny P, Fruscione M, Sloan JA, Schrag D. Symptom Monitoring With Patient-Reported Outcomes During Routine Cancer Treatment: A Randomized Controlled Trial. J Clin Oncol. 2016 Feb 20;34(6):557-65. doi: 10.1200/JCO.2015.63.0830. Epub 2015 Dec 7. PMID 26644527
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org